CLINICAL TRIAL: NCT05466084
Title: A Randomized Controlled Trial Studying Tissue Glue vs Metallic Tackers in Mesh Fixation During TAPP Repair.
Brief Title: Tissue Glue vs Metallic Tackers in Mesh Fixation During TAPP Repair.
Acronym: TAVGLU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jordan (Other)
Responsible Party: Principal Investigator, Hanan Ibrahim Mansour, General surgery specialist, University of Jordan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10/2022/4308
Record Dates: First submitted 2022-07-16; First posted 2022-07-20 (Actual); Last update posted 2022-08-10 (Actual); Status verified 2022-08

CONDITIONS: Hernia
Keywords: Laparoscopic TAPP; tissue glue; tackers; hernia
MeSH Terms: conditions — Hernia

STUDY DESIGN:
Intervention Model Description: randomized control trial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- tissue glue (Experimental): mesh fixed using tissue glue
  Interventions: Procedure: tissue Glue for mesh fixation
- metallic tackers (Experimental): mesh fixed using metallic tackers
  Interventions: Procedure: Metallic Tackers for mesh fixation

INTERVENTIONS:
Procedure: tissue Glue for mesh fixation — one arm of the study had their mesh fixed with tissue glue applied at multiple sites
  Arms: tissue glue
Procedure: Metallic Tackers for mesh fixation — in the other arm mesh was fixed with tackers applied avoiding the triangle of pain and the triangle of doom using a three point fixation technique; Cooper's ligament, medial cranial edge of the mesh and just lateral to the inferior epigastric vessels.
  Arms: metallic tackers

SUMMARY:
This is a randomized control trial intending to study the clinical difference between different mesh fixation techniques in laparoscopic TAPP hernioplasty of inguinal hernia for adults with unilateral and bilateral inguinal hernia , two techniques are tissue glue and surgical tackers , the target population will be divided according to an electronic generated randomization into two groups , they will be compared according to multiple variables which includes but not limited to : procedure time, early post op complication , post-operative pain , late complications , short term and long term recurrence rates .

DETAILED DESCRIPTION:
Laparoscopic transabdominal preperitoneal ( TAPP ) hernioplasty has emerged as an essential procedure for adults complaining of both unilateral and bilateral inguinal hernia , various descriptions of the procedure have been published recently, complications and recurrence rates are being calculated for each method, different mesh fixation techniques are being used by different surgeons, some use surgical tackers, some use fibrin glue and some demonstrated an equal outcome if the mesh was not fixed at all.

This is a randomized control trial intending to study the clinical difference between those different mesh fixation techniques in laparoscopic TAPP hernioplasty of inguinal hernia for adults with unilateral and bilateral inguinal hernia , two techniques are tissue glue and surgical tackers , the target population will be divided according to an electronic generated randomization into two groups , they will be compared according to multiple variables which includes but not limited to : procedure time, early post op complication , post-operative pain , late complications , short term and long term recurrence rates .

ELIGIBILITY:
Inclusion Criteria:

* all Adult Patients ages between 18 and 80 years old, males and females, inguinal hernias, unilateral or bilateral and femoral hernias.

Exclusion Criteria:

* operations which were converted from TAPP to other procedures (such as open repair or TEP).
* Patients who were unfit for general anesthesia
* patients who refused to participate in the study
* patients with chronic pain disorders requiring long term pain management before the procedure.
* cases with complicated hernias that required emergency repair.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
postoperative pain | 6 weeks
  postoperative pain was measured using The visual analog scale ( VAS ) scored from 1-10

SECONDARY OUTCOMES:
postoperative complications | 6 weeks
  postoperative complications including : seroma, ssi , hematoma and others
operative time | intraoperative
  operative time
hospital stay | 6 WEEKS
  postoperative days in hospital measured

CONTACTS AND LOCATIONS:
Locations (1):
- University of Jordan , faculty of medicine, Amman, Jordan

IPD SHARING:
Plan to Share IPD: No